CLINICAL TRIAL: NCT00328263
Title: A Double-blind, Randomized, Placebo Controlled, Multicenter Study of the Efficacy and Safety of BIO-K*+ CL-1285* in the Prevention of Antibiotic-associated Diarrhea in Adult Patients Exposed to Nosocomial Infection.
Brief Title: Efficacy and Safety of BIO-K + CL1285 in Prevention of Antibiotic-associated Diarrhea in Hospitalized Adult Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-K Plus International Inc. (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CL1285-AAD-M01
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Diarrhea; Clostridium Infections
Keywords: Bio-K+CL1285; Probiotics; Antibiotics-associated diarrhea; Clostridium difficile-associated diarrhea; Lactobacillus acidophilus; Clostridium Difficile
MeSH Terms: conditions — Diarrhea; Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Bio-K Cl1285 Bio-K Cl1285 contains 50 billion of live bacteria.
  Interventions: Dietary Supplement: Lactobacillus acidophilus CL1285 and Lactobacillus casei
- 2 (Placebo Comparator): placebo devoid of bacteria
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus acidophilus CL1285 and Lactobacillus casei — One bottle daily 2 hours before or after antibiotic administration and for 5 days following the termination of antibiotic regimen.
  Other Names: BioK CL1285
  Arms: 1
Dietary Supplement: placebo — One bottle daily 2 hours before or after antibiotic administration and for 5 days following the termination of antibiotic regimen.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Bio-K + CL1285 versus placebo in the prevention of antibiotic-associated diarrhea in hospitalized adult patients.

DETAILED DESCRIPTION:
Antibiotic-associated diarrhea (AAD) is one of the most frequent adverse events following antibiotherapy and is the leading cause of diarrhea in hospitalized patients. Ten to 25% of AAD are caused by the bacteria Clostridium difficile.

A recent unicenter study conducted at Maisonneuve-Rosemont hospital demonstrated the preventive role of Bio-K + CL1285 in antibiotic-associated diarrhea and Clostridium difficile-associated diarrhea. Its preventive role is thought to be mainly through restoration of the gastrointestinal flora affected in part by the antibiotherapy.

A wide body of literature reveals clinical use of probiotics, but few well controlled prospective studies conducted on large numbers of subjects have been performed.

In light of the positive preliminary results obtained in a limited number of patients with AAD and of the paucity of well controlled clinical trials, we now wish to undertake a randomized, double blind, multicentre study to evaluate the efficacy and safety of Bio-K + CL1285 prophylaxis vs. placebo in the prevention of antibiotic-associated diarrhea in hospitalized adult patients. As secondary objectives, we also intend to evaluate the incidence of Clostridium difficile-associated diarrhea and to demonstrate that BIO-K + CL1285 agent will not only improve the clinical outcomes but also reduce health care expenditures.

ELIGIBILITY:
Inclusion Criteria:

* presenting to the Emergency Room and considered for admission to hospital for a minimum of 12 hours and requiring antibiotic administration for the treatment of a suspected or proven bacterial infection OR a hospitalized patient developing a suspected or proven nosocomial infection OR an external patient that come to the hospital for repeated visits to receive his intravenous antibiotic therapy for the treatment of a suspected or proven bacterial infection. The external patients on oral antibiotics that come to the hospital for repeated visits to receive any other treatments requiring a hospital stay of more than one hour will also be included.
* Hospital employee on antibiotics can also be included in the study
* having received less than 24 hours of antibiotic therapy;
* requiring a minimum of 3 days and a maximum of 14 days antibiotic administration

Informed consent must be obtained in writing for all subjects at enrollment into the study

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* active diarrhea;
* a history of daily consumption of fermented milk and/or yogurt;
* intolerance to lactose;
* pregnant/breastfeeding women;
* an active, non controlled intestinal disease such as Crohn's Disease or ulcerative colitis;
* ileostomy, jejunostomy or colostomy;
* immunosuppressed state;
* a previous documented C. difficile infection in the three months prior to study initiation;
* active radiotherapy or chemotherapy;
* recent (< 6 months) or planned bone marrow graft or organ transplant;
* antibiotic therapy in the fourteen days prior to study initiation;
* the planned administration of metronidazole (alone or in combination) or vancomycin monotherapy for the treatment of an infection;
* mental or other conditions, or language barriers rendering the subject unable to understand the nature, scope, and possible consequences of the study or complete the self-administered questionnaires;
* subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.

Post-enrollment exclusion criteria include fermented milk and/or yogurt consumption during the study period and two consecutive missed dose of study product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe S Dylewski, MD, Principal Investigator — St-Mary Hospital Center
Locations (8):
- Canada (8):
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - North York General Hospital, Toronto, Ontario
  - Hotel Dieu de Chicoutimi, Chicoutimi, Quebec
  - St-Mary Hospital Center, Montreal, Quebec
  - Laval Hospital, Québec, Quebec
  - Hotel-Dieu de St-Jerome, Saint-Jérôme, Quebec
  - Centre Hospitalier Régional de Trois-Rivières, Trois-Rivières, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2151 patients were screened for eligibility. 437 patients were randomized for the study between March 2006 and October 2006.
Pre-assignment Details: Inclusion & exclusion criterias were used to randomized patients. Patients were followed for an additionnal 21 days after treatment ended.
Groups:
- Bio-K+ CL1285: 98g/day of Bio-K+ CL1285 containing 50 billion of live bacteria.
- Placebo: 98g/day of placebo (devoid of microorganisms)
Period: Overall Study
Arm/Group | Bio-K+ CL1285 | Placebo
Started | 216 | 221
Completed | 213 (3 deaths occured during the study. None of the deaths were causally related to the study product.) | 217 (4 deaths occured during the study. None of the deaths were causally related to the study product.)
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bio-K+ CL1285 | Placebo | Total
Number analyzed (Participants) | 216 | 221 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (18.1) | 58.1 (19.1) | 58.8 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 114 | 213
  Male | 117 | 107 | 224
Region of Enrollment [Number; unit: participants]
  Canada | 216 | 221 | 437

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Antibiotic-associated Diarrhea.
Description: Presence of at least one diarrhea episode within 24 hours.
Time Frame: Up to 40 days
Measure: Number; unit: participants
Arm/Group | Bio-K+ CL1285 | Placebo
Number analyzed (Participants) | 216 | 221
participants | 216 | 221

2. Secondary Outcome: Positive Results for Clostridium Difficile (C. Difficile) Toxin A or B in Antibiotic Associated Diarrhea Patients.
Description: Testing for CDAD was performed at the discretion of the treating physician and according to the protocol in place at the study centers. CDAD was defined as an episode of diarrhea and positive results for C. difficile Toxin A or B.
Time Frame: Up to 40 days
Reporting Status: Not Posted

3. Secondary Outcome: Health Outcome Evaluation Will Look at the Direct Medical Costs and Clinical Outcomes of Alternative Strategies in the Prevention of Antibiotic-associated Diarrhea in Hospitalized Adult Patients
Time Frame: Up to 40 days
Reporting Status: Not Posted

4. Secondary Outcome: Safety Profile of BIO-K+CL1285® Versus Placebo in Patients on Antibiotics
Description: Safety was assessed by the incidence of treatment-emerged adverse events, which were reported according to MedDRA 10.1
Time Frame: Up to 40 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bio-K+ CL1285 | Placebo
Serious Adverse Events (participants affected / at risk) | 15/216 | 23/221
Other Adverse Events (participants affected / at risk) | 109/216 | 113/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bio-K+ CL1285 (N=216) | Placebo (N=221)
Serious Adverse Events (General disorders) | 15 (72) | 23 (76) — None of the serious adverse events were related to the treatment product.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bio-K+ CL1285 (N=216) | Placebo (N=221)
Gastrointestinal adverse events (Gastrointestinal disorders) | 35 | 30 — The most frequently reported non serious adverse events were constipation, flatulence and nausea.
Other adverse events (Nervous system disorders) | 74 | 83 — Vulvovaginal mycotic infection, muscle spasms, hyperthermia, pyrexia, arthralgia, headache, dyspnea, presence of at least one treatment-emergent non serious adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed publication or formal presentation of the data directly derived from the study shall be submitted to Bio-K+. Bio-K+ will have 15 business days to give comments to the Investigator.This review is no way intended to restrict publication of facts or opinions formulated by the Investigator through this research.